CLINICAL TRIAL: NCT05290623
Title: High-power Green-light Laser Endoscopic Submucosal Dissection for Non-muscle-invasive Bladder Cancer: a Technical Improvement and Its Initial Application
Brief Title: High-power Green-light Laser Endoscopic Submucosal Dissection for Non-muscle-invasive Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Muwen Wang, Professor, Shandong Provincial Hospital
Other Study IDs: SWYX:NO. 2022-085
Record Dates: First submitted 2022-03-18; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective study was designed in this study. The surgeon performed high-power green-light laser endoscopic submucosal dissection (HPL-ESD) for the treatment of primary non-muscle-invasive bladder cancer (NMIBC). This surgical treatment was novel and safety and efficacy of the treatment has not been established. We collected relative data in Shandong Provincial Hospital Affiliated to Shandong First Medical University from May 2018 to December 2020. Preoperative, intraoperative and postoperative clinical data were collected and analysed. The safety and efficacy of the novel surgical treatment were verified by the short-term and long-term clinical outcomes. Fifty patients with NMIBC were planed to be enrolled in the study.

DETAILED DESCRIPTION:
Background: In recent years, endoscopic laser surgery has been introduced to the treatment of NMIBC. Various types of laser (holmium laser, thulium laser and green-light laser) have been examined in the treatment of NMIBC, and the cutting power has been raised gradually. In our previous study, a 120 W green-light laser was used to perform en bloc resection, which yielded encouraging results. Endoscopic submucosal dissection by the HybridKnife was reported to be safe and effective in the treatment of NMIBC. However, previous resection was performed by electrical instrument. To further enhance the safety and accuracy of the operation, surgeons improved the treatment by combining laser resection and endoscopic submucosal dissection (ESD). This novel surgical treatment can also integrate advantages of each method. A retrospective study was designed in this study. The aim of the study was to evaluate the safety and efficacy of this novel surgical treatment, high-power green-light laser endoscopic submucosal dissection (HPL-ESD), in the treatment of primary non-muscle-invasive bladder cancer (NMIBC).

Introduction: Greenlight lasers are developed from Nd:YAG laser. Visual laser vaporization with Nd:YAG laser was introduced for the treatment of bladder cancer in the early 1990s. However, the low-absorption in most tissues with a penetration depth of 4-18mm leading to a deep coagulative necrosis of tissue, which increased the risk of delayed bladder perforation and bowel injury. Passing the Nd:YAG-produced beam (1046nm) through a KTP or LBO crystal, leads to a green visible light beam of 532nm, which has a completely different laser beam-tissue interaction. The wavelength is not absorbed by water but strongly absorbed by hemoglobin, which limits the optical penetration depth of green light laser to 0.8 mm, and the heat remaining in the tissue induces a coagulation zone of only 1-2mm thickness. Recent studies show that greenlight laser vaporization is a reliable and feasible treatment for the patients with primary NMIBC compared with standard TURBT.

On the basis of our previous surgical procedure, we developed this new surgical method by introducing ESD technology. Thus LBO laser en bloc resection was combined with the ESD technique to treat NMIBC, which was inspired by waterjet-assisted ESD in the department of gastroenterology. ESD was developed from endoscopic mucosal resection (EMR) and widely applied for the treatment of early gastroesophageal cancer and colorectal neoplasms. The bladder wall shares a similar histological structure with the gastrointestinal tract, although the muscularis propria is thicker. Therefore, forming a submucosal fluid cushion in the bladder wall should be feasible and even safer. The effects of submucosal fluid cushion on bladder wall were showed intuitively. The interspace between the mucosal layer and the detrusor muscle layer was increased, and the tissue between the two layers was rendered looser. In the present study, the submucosal fluid cushion increases safety during the operation. More importantly, when the normal mucosa was incised, the detrusor muscle layer beneath was exposed, which facilitated distinction of which layer was reached and incision of the entire tumor with the superficial detrusor muscle beneath the basal part. To some extent, introduction of the ESD technique enabled safe, controllable and accurate incision.

Equipment: The equipment included a 23F continuous flow resectoscope through which a 6F green-light lithium triborate (LBO) laser fiber (Realton, Beijing, China) could be delivered via the working channel. In addition, a disposable injector was used to form the submucosal fluid cushion for ESD. The stainless steel needle of the injector is 5 mm in length and 0.6 mm in diameter (terminal part). The working length and diameter are 1650 mm and 2.5 mm respectively (middle part), enabling delivery through the working channel of the resectoscope. The beginning part of the injector was connected to a 20-ml syringe containing methylene blue solution as the injection fluid.

HPL-ESD procedure: All surgeries were conducted in the lithotomy position under continuous epidural anesthesia. Sodium chloride physiological solution was used for irrigation. The 23F continuous flow resectoscope was delivered into the bladder through the urethra initially. Each visible tumor was examined to confirm the location, number, and size and the condition of the adjacent mucosa. Then, the 6F green-light LBO laser fiber was delivered through the working channel of the resectoscope. Each tumor was first marked with a circular coagulation blockage border, which was 1-2 cm from the edge of the tumor. Next, the laser fiber was temporarily withdrawn and the disposable injector was delivered through the same working channel of the resectoscope. Multipoint injection was performed in the normal mucosa along the blockage border. Because the tissue between the mucosal layer and the detrusor muscle layer in the bladder wall is relatively loose, a blue submucosal fluid cushion was formed between the two layers after injection. Subsequently, the green-light laser was delivered through the working channel again. The laser power was set at 160 W for cutting and 30-50 W for coagulation simultaneously. The mucosa was incised annularly, and the detrusor muscle layer beneath it was gradually exposed. The submucosal fluid cushion separated the mucosa layer and the detrusor muscle layer to some extent in advance. Therefore, the course and distribution of the detrusor muscle could be clearly observed. Dissection of tissue connected between the tumor and the bladder wall was also facilitated. The entire tumor was excised with superficial detrusor muscle beneath the basal part. After resection, the whole tumor bed and surrounding mucosa were carefully coagulated at a power of 30-50 W. The intact bladder tumor was removed with an alligator forceps or flushed out with an Ellik evacuator. When the tumor size was > 3 cm, the specimen was longitudinally cut into two or more parts.

Clinical data will be collected, such as patient data, tumor characteristics, and perioperative data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-muscle invasive bladder cancer who received high-power green laser submucosal resection of bladder tumor

Exclusion Criteria:

* Patients with muscle invasive bladder cancer
* Patients with recurrent bladder cancer
* Patients with benign bladder tumor

Ages: 20 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary non-muscle invasive bladder cancer that received high-power green laser submucosal resection will be enrolled in this study. Gender is not limited. Most patients were elder male people with smoking history.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Success rate of the surgery | after all data has been collected, analysis will be finished within 5 days
  The success of the surgery was NMIBC got en bloc resection by HPL-ESD without transfering to other treatment. Success rate of the surgery is the proportion of surgery success in all surgery.

SECONDARY OUTCOMES:
Rate of tumor en bloc resection | after all data has been collected, analysis will be finished within 5 days
  The proportion of tumor en bloc resection (R0 resection) in all resected tumors.
Operative time | after all data has been collected, analysis will be finished within 5 days
  The time from the installation of endoscopic instrument to the complete resection of bladder tumor
Hemoglobin decrease | after all data has been collected, analysis will be finished within 5 days
  Hemoglobin decrease (g/dL) = preoperative serum hemoglobin (g/dL) - postoperative serum hemoglobin (g/dL)
Catheterization time | after all data has been collected, analysis will be finished within 5 days
  Time from indwelling catheter intraoperatively to removing catheter postoperatively
Hospital stay | after all data has been collected, analysis will be finished within 5 days
  The hospital stay is the total number of days from the admission to the discharge of patients
Complication | after all data has been collected, analysis will be finished within 5 days
  Obturator nerve reflex, perforation, urethral stricture, hydronephrosis
The recurrence rate of tumor in situ | after all data has been collected, analysis will be finished within 5 days
  The proportion of patients with postoperative tumor recurrence in situ in all patients after a 12-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xishuang S, Deyong Y, Xiangyu C, Tao J, Quanlin L, Hongwei G, Jibin Y, Dongjun W, Zhongzhou H, Jianbo W, Lina W, Lin Y. Comparing the safety and efficiency of conventional monopolar, plasmakinetic, and holmium laser transurethral resection of primary non-muscle invasive bladder cancer. J Endourol. 2010 Jan;24(1):69-73. doi: 10.1089/end.2009.0171. PMID 19954353
- [Background] Zhu Y, Jiang X, Zhang J, Chen W, Shi B, Xu Z. Safety and efficacy of holmium laser resection for primary nonmuscle-invasive bladder cancer versus transurethral electroresection: single-center experience. Urology. 2008 Sep;72(3):608-12. doi: 10.1016/j.urology.2008.05.028. Epub 2008 Jul 23. PMID 18649930
- [Background] Nagele U, Kugler M, Nicklas A, Merseburger AS, Walcher U, Mikuz G, Herrmann TR. Waterjet hydrodissection: first experiences and short-term outcomes of a novel approach to bladder tumor resection. World J Urol. 2011 Aug;29(4):423-7. doi: 10.1007/s00345-011-0653-8. Epub 2011 Feb 9. PMID 21305303
- [Background] Herrmann TR, Wolters M, Kramer MW. Transurethral en bloc resection of nonmuscle invasive bladder cancer: trend or hype. Curr Opin Urol. 2017 Mar;27(2):182-190. doi: 10.1097/MOU.0000000000000377. PMID 28033148
- [Background] Fried NM, Murray KE. High-power thulium fiber laser ablation of urinary tissues at 1.94 microm. J Endourol. 2005 Jan-Feb;19(1):25-31. doi: 10.1089/end.2005.19.25. PMID 15735378
- [Background] He D, Fan J, Wu K, Wang X, Wu D, Li L, Li X, Liu L, Cao P, Cao J, Chang LS. Novel green-light KTP laser en bloc enucleation for nonmuscle-invasive bladder cancer: technique and initial clinical experience. J Endourol. 2014 Aug;28(8):975-9. doi: 10.1089/end.2013.0740. Epub 2014 May 19. PMID 24735433
- [Background] Tao W, Yang D, Shan Y, Xue B, Sun C, Zang Y, Zhang Y. Safety and efficacy of 120W high performance system greenlight laser vaporization for non-muscle-invasive bladder cancer. J Xray Sci Technol. 2013;21(2):309-16. doi: 10.3233/XST-130379. PMID 23694918
- [Background] Bai Y, Liu L, Yuan H, Li J, Tang Y, Pu C, Han P. Safety and efficacy of transurethral laser therapy for bladder cancer: a systematic review and meta-analysis. World J Surg Oncol. 2014 Sep 25;12:301. doi: 10.1186/1477-7819-12-301. PMID 25256383
- [Background] Chen J, Zhao Y, Wang S, Jin X, Sun P, Zhang L, Wang M. Green-light laser en bloc resection for primary non-muscle-invasive bladder tumor versus transurethral electroresection: A prospective, nonrandomized two-center trial with 36-month follow-up. Lasers Surg Med. 2016 Nov;48(9):859-865. doi: 10.1002/lsm.22565. Epub 2016 Jul 25. PMID 27454755
- [Background] Kramer MW, Rassweiler JJ, Klein J, Martov A, Baykov N, Lusuardi L, Janetschek G, Hurle R, Wolters M, Abbas M, von Klot CA, Leitenberger A, Riedl M, Nagele U, Merseburger AS, Kuczyk MA, Babjuk M, Herrmann TR. En bloc resection of urothelium carcinoma of the bladder (EBRUC): a European multicenter study to compare safety, efficacy, and outcome of laser and electrical en bloc transurethral resection of bladder tumor. World J Urol. 2015 Dec;33(12):1937-43. doi: 10.1007/s00345-015-1568-6. Epub 2015 Apr 25. PMID 25910478
- [Background] Lingenfelder T, Fischer K, Sold MG, Post S, Enderle MD, Kaehler GF. Combination of water-jet dissection and needle-knife as a hybrid knife simplifies endoscopic submucosal dissection. Surg Endosc. 2009 Jul;23(7):1531-5. doi: 10.1007/s00464-009-0433-3. Epub 2009 Apr 3. PMID 19343433
- [Background] Park JS, Youn YH, Park JJ, Kim JH, Park H. Clinical Outcomes of Endoscopic Submucosal Dissection for Superficial Esophageal Squamous Neoplasms. Clin Endosc. 2016 Mar;49(2):168-75. doi: 10.5946/ce.2015.080. Epub 2016 Feb 12. PMID 26867548
- [Background] Cheng YY, Sun Y, Li J, Liang L, Zou TJ, Qu WX, Jiang YZ, Ren W, Du C, Du SK, Zhao WC. Transurethral endoscopic submucosal en bloc dissection for nonmuscle invasive bladder cancer: A comparison study of HybridKnife-assisted versus conventional dissection technique. J Cancer Res Ther. 2018;14(7):1606-1612. doi: 10.4103/jcrt.JCRT_786_17. PMID 30589047
- [Background] Fritsche HM, Otto W, Eder F, Hofstadter F, Denzinger S, Chaussy CG, Stief C, Wieland WF, Burger M. Water-jet-aided transurethral dissection of urothelial carcinoma: a prospective clinical study. J Endourol. 2011 Oct;25(10):1599-603. doi: 10.1089/end.2011.0042. Epub 2011 Aug 4. PMID 21815824
- [Background] Kaehler GF, Sold MG, Fischer K, Post S, Enderle M. Selective fluid cushion in the submucosal layer by water jet: advantage for endoscopic mucosal resection. Eur Surg Res. 2007;39(2):93-7. doi: 10.1159/000099597. Epub 2007 Feb 13. PMID 17299266
- [Background] Xu Y, Guan W, Chen W, Xie C, Ouyang Y, Wu Y, Liu C. Comparing the treatment outcomes of potassium-titanyl-phosphate laser vaporization and transurethral electroresection for primary nonmuscle-invasive bladder cancer: A prospective, randomized study. Lasers Surg Med. 2015 Apr;47(4):306-11. doi: 10.1002/lsm.22342. Epub 2015 Apr 9. PMID 25864416